CLINICAL TRIAL: NCT02667561
Title: Phase I Clinical Trial for Evaluation of Pharmacokinetics, Pharmacodynamics and Safety of Testosterone Gel 1% for Topical Use, After Administration of Three Different Doses (2.2 mg, 4.4 mg, 8.8 mg and Placebo) for 28 Consecutive Days in Post-menopausal Women.
Brief Title: Pharmacokinetics, Pharmacodinamic and Safety of Testosterone Gel 1%
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study has been cancelled and it has not been initiated.
Sponsor: Biolab Sanus Farmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GDN 060/15
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2017-09

CONDITIONS: Post-menopausal Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Testosterone gel 1% 2.2 mg (Experimental): Testosterone gel 1% Topical use 2.2 mg (220 mg of gel) once daily duration of treatment: 28 days
  Interventions: Drug: Testosterone gel 1% 2.2 mg
- Testosterone gel 1% 4.4 mg (Experimental): Testosterone gel 1% Topical use 4.4 mg (440 mg of gel) once daily duration of treatment: 28 days
  Interventions: Drug: Testosterone gel 1% 4.4 mg
- Testosterone gel 1% 8.8 mg (Experimental): Testosterone gel 1% Topical use 8.8 mg (880 mg of gel) once daily duration of treatment: 28 days
  Interventions: Drug: Testosterone gel 1% 8.8 mg
- Placebo of Testosterone Gel 1% (Placebo Comparator): Placebo of Testosterone Gel 1% Topical use Approximately 550 mg of gel Once daily duration of treatment: 28 days
  Interventions: Drug: Placebo of Testosterone Gel 1%

INTERVENTIONS:
Drug: Testosterone gel 1% 2.2 mg — Application of 220 mg of Testosterone Gel 1% in pubic region, once daily, for 28 consecutive days.
  Arms: Testosterone gel 1% 2.2 mg
Drug: Testosterone gel 1% 4.4 mg — Application of 440 mg of Testosterone Gel 1% in pubic region, once daily, for 28 consecutive days.
  Arms: Testosterone gel 1% 4.4 mg
Drug: Testosterone gel 1% 8.8 mg — Application of 880 mg of Testosterone Gel 1% in pubic region, once daily, for 28 consecutive days.
  Arms: Testosterone gel 1% 8.8 mg
Drug: Placebo of Testosterone Gel 1% — Application of approximately 550 mg of Placebo of Testosterone Gel 1% in pubic region, once daily, for 28 consecutive days.
  Arms: Placebo of Testosterone Gel 1%

SUMMARY:
This is a Phase I, open-label, parallel trial to evaluate Pharmacokinetics, Pharmacodynamics and Safety of Testosterone gel 1% for topic usage in post-menopausal women, for 28 days

DETAILED DESCRIPTION:
This is a Phase I, open-label, parallel trial to evaluate Pharmacokinetics, Pharmacodynamics and Safety of Testosterone gel 1% for topic usage in post-menopausal women, Study participants will receive investigational product for 28 consecutive days, once daily, as per the following allocation: 2.2 mg, 4.4 mg. 8.8 mg or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged ≥ 42 years and ≤ 65 years, in post-menopausal period for at least 1 year and with active sexual life;
* Serum testosterone levels < 33 ng/mL;
* Follicle-stimulating hormone (FSH) levels > 22 mU/mL;
* Absence of other significant diseases which, at the physician's discretion, could impact subject's participation in the trial, according to protocol requirements, and study evaluations: medical history, blood pressure and heart rate measurements, physical examination and complimentary laboratory tests;
* Ability to understand the nature and objective of the trial, including risks and adverse events, which shall be confirmed by Informed Consent Form signature.

Exclusion Criteria:

* Screening laboratory tests results presenting clinically relevant deviations that, at the investigator discretion, prevent the subject to participate in the trial due to possible risks;
* Drugs addiction, including alcohol;
* Treatment with any drugs known to have a well-established toxic potential to major organs, within 3 months before the trial, ;
* Participation in any other experimental research or administration of any experimental drug within six months before the initiation of this trial;
* Pregnancy, labor or miscarriage in the last 12 weeks before the antecipated date of the study treatment start;
* Any conditions, according to investigator's best judgement, that prevents the subject to participate in the trial.

Ages: 42 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics, area under the curve (AUC) | 28 days
Pharmacokinetics, maximum concentration (Cmax) | 28 days
Pharmacokinetics, time to maximum concentration (Tmax) | 28 days
Pharmacokinetics, half-life (t1/2) | 28 days

SECONDARY OUTCOMES:
Pharmacodynamics, response rate, by Female Sexual Function Index | 28 days
Safety, number of adverse events | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto De Nucci, PhD, Principal Investigator — Galeno Desenvolvimento de Pesquisas

IPD SHARING:
Plan to Share IPD: No